CLINICAL TRIAL: NCT04859153
Title: Relevant Factors on Sprint Performance in Adolescent Sprinters: Influences of Central Visuomotor and Audiomotor Mechanisms, Muscle Mechanical Properties and Skill-related Physical Fitness
Brief Title: Relevant Factors on Sprint Performance in Adolescent Sprinters
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRREC-109-195
Record Dates: First submitted 2021-03-28; First posted 2021-04-26 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Sprint Performance; Physical Fitness; Muscle Architecture; Reaction Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sprinter: All sex of healthy adolescent athletes of the athletics sprint
  Interventions: Diagnostic Test: central nerve sensory, motor control and various muscle mechanical characteristic and sport-related fitness test
- Non-sprinter: All sex of healthy adolescent athletes of other kinds of sports
  Interventions: Diagnostic Test: central nerve sensory, motor control and various muscle mechanical characteristic and sport-related fitness test

INTERVENTIONS:
Diagnostic Test: central nerve sensory, motor control and various muscle mechanical characteristic and sport-related fitness test — To explore the sports performance of the adolescent sprinters, including analyzing the correlations between the results and central nerve sensory, and also between motor control and various muscle mechanical characteristic and sport-related fitness factor.

SUMMARY:
Purpose: To explore the sports performance of the adolescent sprinters, including analyzing the correlations between the results and central nerve sensory, and also between motor control and various muscle mechanical characteristic and sport-related fitness factor.

DETAILED DESCRIPTION:
The sprint performance was determined by various relevant factors, and they were mainly divided into central system factor and peripheral system factor. An effective sprint start requires a quick reaction to an auditory stimulus followed by a determined sequence of activation of particular muscles responsible for maximum movement speed. Both of the skill-related physical fitness, including muscle strength, muscle endurance, muscle power, speed, agility, and balance, and muscle physical characteristic, including muscle tone and muscle architecture, are related to the sprint performance. The 100m race could divided into three different phases, start acceleration, maximum speed, and deceleration. According to Collet, 1999, the determinants of the temporal structure of the sprint start are RT, movement speed and movement frequency, which involves in perfecting sprinters' physical performance. And also, according to Pilianidis et al., 2012; Tonnessen et al., 2013, the start reaction time significantly affects the reduction of running time in 100 m races. In the recent studies, there are researches only showing that the auditory stimulus trainings significantly affected the final results for swimming athletes, and that the visual stimulus trainings significantly affected the final scores for badminton athletes.This study will mainly recruit the healthy adolescent athletes of the athletics sprint and other kinds of sports in the age range 13-18 years, and will evaluate the athletes of anthropometric measurements and physical fitness, 100m sprint performance, muscle characteristic, jump ability, agility, and nerve potential measurements.The outcome of this study will be able to be one of the comprehensive trials for coaches to take into consideration when choosing their own athletes. And also, the athletes may choose their own specialties that fit their own physical conditions. Moreover, the adolescent athletes will be trained more precisely and effectively. These will positively lead to reaching their personal best results and decreasing the occurrences of the sport injuries due to unsuitable events and trainings.

ELIGIBILITY:
Inclusion Criteria:

* the healthy adolescent athletes of the athletics sprint and other kinds of sports

Exclusion Criteria:

* cardiovascular diseases
* lower extremities surgery histories
* musculoskeletal sports injuries that would affect the sports testing
* auditory or visual disabilities
* brain injury histories.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the healthy adolescent athletes of the athletics sprint and other kinds of sports
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Distance of vertical jump.horizontal jump and hexagonal barbell jump squat | day 1
  Use data collection sensor (Vmaxpro, Germany) to measure.
  * vertical jump :; The subject will in an upright posture when preparing for the action. At the beginning, they will squat down until knees were bent 90 degrees, and jump as high as possible.
  * horizontal jump : The subject's leg should be shoulder-width apart, squat and jump forward as far as possible.
  * hexagonal barbell jump squat : The subject will perform five different weight jumps (0%, 10%, 20%, 30% and 40% of 1RM) with a 15 kg hexagonal barbell, they will squat down until knees were bent 90 degrees, and jump as high as possible.
  The data collection sensor will detect the highest and farthest distance(meters).
Power of vertical jump.horizontal jump and hexagonal barbell jump squat | day 1
  Use data collection sensor (Vmaxpro, Germany) to measure.
  * vertical jump : The subject will in an upright posture when preparing for the action. At the beginning, they will squat down until knees were bent 90 degrees, and jump as high as possible.
  * horizontal jump : The subject's leg should be shoulder-width apart, squat and jump forward as far as possible.
  * hexagonal barbell jump squat : The subject will perform five different weight jumps (0%, 10%, 20%, 30% and 40% of 1RM) with a 15 kg hexagonal barbell, they will squat down until knees were bent 90 degrees, and jump as high as possible.
  The data collection sensor will detect the velocity and time and use the following formula to calculate the power.
  P=power(W), F=force(kg*m/s^2), V=velocity(m/s),a= acceleration(m/s^2), M=body mass(kg), D= displacement(meters), T=time(seconds)
  * P=F*V(kg*m^2/s^3)
  * F=M*a(kg*m/s^2)
  * V=D/T(m/s)
T-test | day 1
  To measure agility.Set a T-shape with cones. The subject starts from the starting line and starts timing. The subject sprints forward 10 meters to touches the cone A, and then sprints runs to the right for 5 meters to touches the cone B, then move 10 meters to the left and touches the cone C. Finally, move to the right to touches the cone A, then run back across the finish line. Stopped timing when subject passed the finish line. Redcord the best result (seconds).
Hexagonal Obstacle Test | day 1
  To measure agility. Stick a hexagon with a side length of 66 cm on the ground with black tape. The subject's starting position is in the middle of the hexagon. After starting the timing, jump out of each side in order, and then return to the starting position. Stopped timing when after the subject returns to the starting position. Redcord the best result (seconds).
Thickness of muscle | day 1
  Using the liner transducer, 5M-Hz, B(brightness)-mode. The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows muscle thickness(centimeter) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Pennation angle of muscle | day 1
  Using the liner transducer, 5M-Hz, B(brightness)-mode. The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows pennation angle (degree) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Fascicle length of muscle | day 1
  Using the liner transducer, 5M-Hz, B(brightness)-mode. The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows fascicle length (centimeter) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Muscle tone | day 1
  Using the hand-held device MyotonPRO The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows muscle tone(Hz) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Muscle stiffness | day 1
  Using the hand-held device MyotonPRO The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows muscle stiffness (N/m) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Muscle elasticity | day 1
  Using the hand-held device MyotonPRO The measurement of the knee extensor muscle is located midway between the anterior superior iliac spine and the superior part of the patella.
  The measurement of the knee flexor muscle is located midway between the ischial tuberosity and the lateral epicondyle of the tibia.
  The measurement of the plantarflexor muscle is located at the proximal 30% between the lateral malleolus and the lateral condyle of the tibia.
  It shows muscle elasticity (Decrement) of the knee extensor muscle, knee flexor muscle and plantarflexor muscle.
Visuomotor reaction time | day 1
  Measure visual reaction time by Electroencephalography(EEG) Use Neurosoft 21 channel upgradeable EEG system (Neurosoft Neuron Spectrum 4, Russia) to collect EEG data.The electrodes will be put on with plastic caps and distributed evenly on both sides of the brain. The electrical reference will be affixed to O1, O2 and AFz.
  The subject must respond to slow motion onset visual stimulus. When the subject sees the moving visual stimulus on the screen, press the designated button with the index finger of the dominant hand at the fastest speed and the shortest time. The two stimuli will be randomly separated by 2-6 seconds.
  The EEG will show alpha waves include frequency, amplitude, waveform and time of reaction time.
Audiomotor reaction time | day 1
  Measure auditory reaction time by Electroencephalography(EEG) Use Neurosoft 21 channel upgradeable EEG system (Neurosoft Neuron Spectrum 4, Russia) to collect EEG data.The electrodes will be put on with plastic caps and distributed evenly on both sides of the brain. The electrical reference will be affixed to FCz and AFz.
  The subject must respond to slow motion onset auditory stimulus. When hearing the auditory stimulus, the subject must use the index finger of the dominant hand to press the designated button at the fastest speed and the shortest time. There will be a random interval of 2-6 seconds between the two stimuli.
  The EEG will show alpha waves include frequency, amplitude, waveform and time of reaction time.
100 meter sprint performance | day 1
  An light gate was used to measure the subjects' 100m sprint performance. Two light gate were placed at the starting line and the finish line. There were 2 tests in total. The best result (second) was selected for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jia -Min Wu, Principal Investigator — Yueh-Ling Hsieh's graduate student
Locations (1):
- Yueh - Ling Hsieh, Taichung, Taiwan